CLINICAL TRIAL: NCT03363815
Title: A Phase 1, Four-part, Fixed-sequence, Open-label Study to Evaluate the Effect of Multiple Doses of CC-90001 on the Pharmacokinetics of Omeprazole, Midazolam, Warfarin, Rosuvastatin, Metformin, Digoxin, and Nintedanib in Healthy Adult Subjects
Brief Title: A Study to Evaluate the Effect of Multiple Doses of CC-90001 on the Pharmacokinetics of Omeprazole, Midazolam, Warfarin, Rosuvastatin, Metformin, Digoxin, and Nintedanib in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CC-90001-CP-004; U1111-1205-5329 (Registry Identifier: WHO)
Record Dates: First submitted 2017-12-01; First posted 2017-12-06 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Heathy Volunteer
Keywords: Healthy Volunteer; CC-90001; Pharmacokinetics; Omeprazole; Midazolam; Warfarin; Rosuvastatin; Metformin; Digoxin; Nintedanib
MeSH Terms: interventions — CC-90001; Omeprazole; Midazolam; Warfarin; Vitamin K; Rosuvastatin Calcium; Metformin; Digoxin; nintedanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part1:Omeprazole + Midazolam + Warfarin + Vitamin K + CC-90001 (Experimental): Patient will receive CC-90001, 20mg Omeprazole, 2mg Midazolam 10mg Warfarin and 10mg Vitamin K
  Interventions: Drug: CC-90001; Drug: Omeprazole; Drug: Midazolam; Drug: Warfarin; Dietary Supplement: Vitamin K
- Part 2- Rosuvastatin and CC-90001 (Experimental): Patients will receive CC-90001 and 10mg of Rosuvastatin
  Interventions: Drug: CC-90001; Drug: Rosuvastatin
- Part 3: Metformin + Digoxin and CC-90001 (Experimental): Patients will receive CC-90001, 500mg Metformin and 0.25mg, Digoxin
  Interventions: Drug: CC-90001; Drug: Metformin; Drug: Digoxin
- Part 4: Nintedanib and CC-90001 (Experimental): Patients will receive CC-90001 and 100mg of Nintedanib
  Interventions: Drug: CC-90001; Drug: Nintedanib

INTERVENTIONS:
Drug: CC-90001 — CC-90001
Drug: Omeprazole — Omeprazole
  Arms: Part1:Omeprazole + Midazolam + Warfarin + Vitamin K + CC-90001
Drug: Midazolam — Midazolam
  Arms: Part1:Omeprazole + Midazolam + Warfarin + Vitamin K + CC-90001
Drug: Warfarin — Warfarin
  Arms: Part1:Omeprazole + Midazolam + Warfarin + Vitamin K + CC-90001
Dietary Supplement: Vitamin K — Vitamin K
  Arms: Part1:Omeprazole + Midazolam + Warfarin + Vitamin K + CC-90001
Drug: Rosuvastatin — Rosuvastatin
  Arms: Part 2- Rosuvastatin and CC-90001
Drug: Metformin — Metformin
  Arms: Part 3: Metformin + Digoxin and CC-90001
Drug: Digoxin — Digoxin
  Arms: Part 3: Metformin + Digoxin and CC-90001
Drug: Nintedanib — Nintedanib
  Arms: Part 4: Nintedanib and CC-90001

SUMMARY:
This is a four-part study to evaluate the effect of multiple doses of CC-90001 on the PK, safety, and tolerability of single doses of omeprazole, midazolam, warfarin, rosuvastatin, metformin, digoxin, and nintedanib in healthy subjects. Each study part is a nonrandomized, fixed-sequence, open-label, two-period study. The study parts can be run in any order and can be, but do not have to be, run in parallel. Subjects may participate in one part only. For each part, each subject will participate as follows:

* Screening (Days -21 through -2)
* Baseline phase for each study period (Periods 1 and 2)
* Treatment phase for each study period (Periods 1 and 2)
* Follow-up telephone call

DETAILED DESCRIPTION:
This study will consist of 4 parts. Each part has two periods. The parts may be conducted in any order. Subjects may participate in 1 part only.

Each subject will participate in a screening phase, a baseline phase in each study period, a treatment phase in each study period and a follow-up telephone call. Subjects will be screened for eligibility. Eligible subjects will return to the study center on Day -1 of Period 1 and will remain at the study center until the last day of Period 2.

In Part 1, Single doses of omeprazole, midazolam, warfarin, and vitamin K will be administered under fasted conditions on Period 1, Day 1. During Period 2, subjects will receive once daily (QD) doses of CC-90001 from Days 1 through 18. On the day of dosing with probe drugs, CC-90001 will be dosed following an overnight fast. On all other days, CC-90001 can be dosed without regard to food. On Period 2, Day 14, subjects will also be administered single doses of omeprazole, midazolam, warfarin, and vitamin K under fasted conditions.

In Part 2, A single dose of rosuvastatin will be administered under fasted conditions on Period 1, Day 1. There will be a washout period of 5 to 10 days between Period 1, Day 1 and Period 2, Day 1. During Period 2, subjects will receive QD doses of CC-90001 from Days 1 through 6. On the day of dosing with probe drug, CC-90001 will be dosed following an overnight fast. On all other days, CC 90001 can be dosed without regard to food. On Period 2, Day 5, subjects will also be administered a single dose of rosuvastatin under fasted conditions.

In Part 3, single doses of metformin and digoxin will be administered under fasted conditions on Period 1, Day 1.

There will be a washout period of 5 to 10 days between Period 1, Day 1 and Period 2, Day 1. During Period 2, subjects will receive QD doses of CC-90001 from Days 1 through 6. On the day of dosing with probe drugs, CC-90001 will be dosed following an overnight fast. On all other days, CC 90001 can be dosed without regard to food. On Period 2, Day 5, subjects will also be administered single doses of metformin and digoxin under fasted conditions.

In Part 4, a single dose of nintedanib will be administered 30 minutes after the start of a standard breakfast on Period 1, Day 1. There will be a washout period of 5 to 10 days between Period 1, Day 1 and Period 2, Day 1. During Period 2, subjects will receive QD doses of CC-90001 from Days 1 through 14. On the day of dosing with probe drug, CC 90001 will be dosed 30 minutes after the start of a standard breakfast. On all other days, CC 90001 can be dosed without regard to food. On Period 2, Day 14, subjects will also be administered a single dose of nintedanib 30 minutes after the start of a standard breakfast.

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy all of the following criteria to be eligible for enrollment into the study:

* Must understand and voluntarily sign a written informed consent form (ICF) prior to any study-related assessments/procedures being performed.
* Must be able to communicate with the investigator and to understand and adhere to the study visit schedule and other protocol requirements.
* Must be a male or female of any race, aged ≥ 18 to ≤ 64 years of age (inclusive) at the time of signing the ICF.
* Females of childbearing potential (FCBP) must agree to ongoing pregnancy testing during the course of the study and at the end of the study. This applies even if the subject practices true abstinence from heterosexual contact. Note: Females of childbearing potential are not permitted in Part 4.
* Part 4 only: Female subjects must be of nonchildbearing potential as confirmed by medical history. Females of childbearing potential are permitted in Parts 1, 2, and 3.
* Male subjects must practice true abstinence from heterosexual contact (which must be reviewed on a monthly basis, as applicable) or agree to use a male condom (latex or nonlatex condom not made out of natural [animal] membrane [eg, polyurethane]) during sexual contact with a pregnant female or a FCBP while participating in the study and for at least 28 days after the last dose of study drug, even if he has undergone a successful vasectomy as confirmed by medical history.
* Must have a body mass index ≥ 18 and ≤ 33 kg/m2 (inclusive) at the time of signing the ICF.
* Must be healthy as determined by the investigator on the basis of medical history, clinical laboratory test results, vital signs, and 12-lead ECG at screening and Period 1 check-in, as applicable:
* Must be afebrile (febrile is defined as ≥ 38°C or 100.3°F).
* Systolic blood pressure must be in the range of 90 to 140 mmHg, diastolic blood pressure must be in the range of 55 to 90 mmHg, and pulse rate must be in the range of 50 to 110 bpm. Repeat vital signs may be measured at investigator discretion.
* Corrected QT interval using Fridericia's formula (QTcF) value must be ≤ 430 msec for male subjects and ≤ 450 msec for female subjects. An ECG may be repeated up to two times, and the average of the QTcF values will be used to determine subject eligibility.

Exclusion Criteria:

The presence of any of the following will exclude a subject from enrollment into the study:

* History (ie, within 3 years) of any clinically significant neurological, gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, endocrine, hematological, dermatological, psychological, or other major disorders as determined by the investigator.
* Any condition, including the presence of laboratory abnormalities, that places the subject at unacceptable risk if he or she were to participate in the study or confounds the ability to interpret data from the study (congenital nonhemolytic hyperbilirubinemia [eg, Gilbert's syndrome] is not acceptable).
* Use of any prescribed systemic or topical medication, including vaccines, within 30 days of the first dose administration.
* Use of any nonprescribed systemic or topical medication (including vitamin/mineral supplements and herbal medicines) within 14 days of the first dose administration.
* Use of any metabolic enzyme inhibitors or inducers that would affect the relevant drugs for that part of the study within 30 days of the first dose administration unless determined by the investigator that there will be no impact on the study integrity or subject safety. The Indiana University "P450 Drug Interaction Table" should be used to determine inhibitors and/or inducers of metabolic enzymes (http://medicine.iupui.edu/clinpharm/ddis/table/aspx).
* Exposure to an investigational drug (new chemical entity) within 30 days preceding the first dose administration or 5 half-lives of that investigational drug, if known (whichever is longer).
* Presence of any surgical or medical conditions possibly affecting drug absorption, distribution, metabolism, and excretion (eg, bariatric procedure). Appendectomy and cholecystectomy are acceptable.
* Donated blood or plasma within 8 weeks before the first dose administration.
* History of drug abuse (as defined by the current version of the Diagnostic and Statistical Manual [DSM]) within 2 years before dosing or positive drug screening test reflecting consumption of illicit drugs.
* History of alcohol abuse (as defined by the current version of the DSM) within 2 years before dosing or positive alcohol screen.
* Known to have serum hepatitis; known to be a carrier of the hepatitis B surface antigen (HBsAg), hepatitis B surface antibody (anti-HBs), hepatitis B core antibody (anti-HBc), or hepatitis C antibody (HCV Ab); have a positive result to the test for hepatitis B or hepatitis C virus at screening or have a positive result to the test for human immunodeficiency virus (HIV) antibodies at screening. Subjects whose results are compatible with prior immunization against hepatitis B may be included at the discretion of the investigator.
* Use of tobacco- or nicotine-containing products within 3 months prior to Period 1 check in.
* History of multiple drug allergies (ie, 2 or more).
* Are allergic to or hypersensitive to any of the drugs used in the part of the study in which the subject will participate.
* Has any medical condition, medical history, or concomitant medication that is contraindicated in the applicable drug labeling.
* Female subject who is pregnant or breastfeeding. Part 4 only: Female of childbearing potential.
* Additional criteria for Part 1 only:
* History of any significant head trauma as determined by the investigator.
* History of major surgery within 3 months of screening or planned surgery within 14 days of the last dose of study drug.
* Any clinically significant current evidence, personal history, or family history of disorder of hemostasis, congenital or acquired bleeding tendency, or thrombocytopenia.
* History of hemorrhagic diathesis, bleeding complication after surgical procedure or trauma, nose or gingival bleeding, gastrointestinal ulcers with hemorrhage, or menorrhagia (females only).

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2017-12-04 (Actual); Primary Completion 2018-07-29 (Actual); Study Completion 2018-07-29 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic- Cmax | up to approximately 2.5 months
  Maximum observed plasma concentration
Pharmacokinetic- AUC0-t | up to approximately 2.5 months
  AUC from time zero to the last quantifiable concentration

SECONDARY OUTCOMES:
Adverse Events (AEs) | From enrollment until at least 28 days after completion of study treatment
  Number of participants with adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Ramirez-Valle, MD, PhD., Study Director — Celgene
Locations (1):
- Covance Clinical Research Unit, Daytona Beach, Florida, United States